CLINICAL TRIAL: NCT04942197
Title: Evaluation of Fetal Realization Service Using Fetal 3D Avatar Creation and Health Care Application for Pregnant Women
Brief Title: Fetal 3D Avatar Creation for Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: B-2106/688-302
Record Dates: First submitted 2021-06-25; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Virtual Reality; Pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants who received three dimensional ultrasound with pregnancy application
  Interventions: Other: use pregnancy management application
- Arm 2 (Placebo Comparator): Participants who received three dimensional ultrasound without pregnancy management application
  Interventions: Other: use pregnancy management application

INTERVENTIONS:
Other: use pregnancy management application — Pregnant women who used pregnancy management application, which tells patients what she need to know during pregnancy, when to perform tests, and what precautions to take for your baby.

SUMMARY:
* Pregnant women can intuitively check the shape and development of the fetus through the 3D avatar that reflects the characteristics of the fetus. Through a survey on VR fetal experience content and 3D fetal avatar service, the satisfaction of pregnant women/guardians, the bond between the fetus and the mother, and Assess the degree of maternal anxiety.
* Evaluate whether it can be helpful in prenatal monitoring of pregnant women through the use of maternity health management applications, and improve understanding of fetal growth and development.

DETAILED DESCRIPTION:
* This study is an extension of the prospective pilot study conducted in 2020 under the title of "Development of 3D fetal avatar generation technology and fetal experience service technology reflecting the characteristics of pregnant women". In a previous study, about 80% of the mothers who responded to the questionnaire about the similarity of the avatar's fetal face gave a positive answer. Therefore, the developed 3D avatar fetal feeling technology is expected to have a positive effect on the intimacy between the mother and the fetus. want to analyze Pre-developed VR technology is provided through randomization to mothers who have agreed to participate in the study. In addition, objective comparison of prenatal care indicators is provided to mothers who wish to participate in this study by providing a prenatal management application that can comprehensively manage blood pressure, blood sugar, diet, exercise, maternal weight, medications, and expected fetal weight. We intend to evaluate the evaluation and maternal satisfaction.
* If technology and services for simulating a fetus with a 3D fetal avatar are provided, mothers can obtain information such as the face and developmental status of the fetus specialized for their fetus through the 3D fetal avatar. In addition, providing a fetal heart rate simulation linked to the fetal heart sound improves the bond between the mother and the fetus, which can have a positive effect on health, as well as reducing depression during pregnancy and postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women receiving outpatient treatment at Seoul National University Bundang Hospital and pregnant women in the obstetrics and gynecology ward who wish to participate in this study

Exclusion Criteria:

* If Pregnant women refuse to participate in this study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes after using the pregnant woman application | 1 month after examination
  After 3D ultrasonography, at least 1 month later, a questionnaire about bonding between mother and fetus/maternal depression/health management is conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeong-gi Do, South Korea

IPD SHARING:
Plan to Share IPD: No
There are no plans to disclose the records of mothers participating in the study.

REFERENCES:
- [Derived] Lee KN, Kim HJ, Choe K, Cho A, Kim B, Seo J, Myung W, Park JY, Oh KJ. Effects of Fetal Images Produced in Virtual Reality on Maternal-Fetal Attachment: Randomized Controlled Trial. J Med Internet Res. 2023 Feb 24;25:e43634. doi: 10.2196/43634. PMID 36826976